CLINICAL TRIAL: NCT00660712
Title: Evaluation of Patient Characteristics and Treatment Approaches to Patients With Bipolar Disorder in Turkey
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Other Study IDs: NIS-NTR-DUM-2007/1
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; patient characteristics; treatment characteristics
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with bipolar disorder

SUMMARY:
A registry study to identify the patient-diagnosis-treatment characteristic profile of patients with bipolar disorder in Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously or currently diagnosed with bipolar disorder
* Patients (or any of their relatives) who give a written informed consent.

Exclusion Criteria:

* Patients who were previously included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Speciality care outpatient clinic (Psychiatry outpatient clinic)
Sampling Method: Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2008-03; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Identification of the patient-diagnosis-treatment characteristic profile of patients with bipolar disorder in Turkey.

SECONDARY OUTCOMES:
Evaluation of the time period that elapsed since the diagnosis of bipolar disorder
Evaluation of co-morbid psychiatric diseases
Identification of treatment modalities selected according to the disease phase
Identification of the number of first degree relatives diagnosed with bipolar disorder
Evaluation of the relationship between patient and disease characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Bilici, MD, Assoc. Prof, Study Director — Erenkoy State Hospital for Psychiatric Diseases, Istanbul, Turkey
Locations (19):
- Turkey (Türkiye) (19):
  - Research Site, Adana
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Aydin
  - Research Site, Batman
  - Research Site, Denizli
  - Research Site, Erzincan
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Konya
  - Research Site, Malatya
  - Research Site, Mardin
  - Research Site, Mersin
  - Research Site, Rize
  - Research Site, Samsun
  - Research Site, Sivas
  - Research Site, Trabzon